CLINICAL TRIAL: NCT03034577
Title: A Randomized Trial of Deep Neuromuscular Blockade Reversed With Sugammadex Versus Moderate Neuromuscular Block Reversed With Neostigmine, on Postoperative Quality of Recovery
Brief Title: Deep Neuromuscular Block for Laparoscopic Surgery
Acronym: DEEPBLOCK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Melbourne Health (Other); Peter MacCallum Cancer Centre, Australia (Other); Royal Hospital For Women (Other); Northpark Private Hospital (Unknown)
Responsible Party: Principal Investigator, Colin Royse, Professor of Anesthesia, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016.343
Record Dates: First submitted 2017-01-17; First posted 2017-01-27 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Laparoscopy; Anesthesia Recovery Period
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ModNMB (Active Comparator): Moderate Neuromuscular block: participants will receive moderate neuromuscular blockade with rocuronium aiming for TOF 0-2 twitches, with neostigmine reversal when the TOF at least 3 twitches. The depth of neuromuscular block may be reduced after completion of the majority of surgical excision to TOF 3 or more
  Neostigmine
  Interventions: Drug: Neostigmine
- DeepNB (Active Comparator): Deep Neuromuscular block: participants will receive DNB aiming for a post tetanic count of 1-2, which will be maintained until removal of the laparoscopic ports, with reversal using sugammadex
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — Reversal of neuromuscular block Sugammadex dosage will be adjusted to body weight and PTC/TOF count at the time of reversal, and not administered until PTC at least 1. Dosage will be 4mg/kg if TOF = 0 and PTC ≥ 1; and 2 mg/kg if TOF ≥1.
  Arms: DeepNB
Drug: Neostigmine — Neostigmine 50 micrograms/kg coupled with atropine 20 micrograms/kg or glycopyrrolate 5 micrograms/kg, to a maximum dose of neostigmine of 5.0 mg. The neostigmine should not be administered until the TOF has at least 3 twitches present.
  Arms: ModNMB

SUMMARY:
Trial summary: deep neuromuscular block is proposed as a technique to improve operative conditions for laparoscopy. Early clinical data would suggest that there may also be patient benefits beyond the operative period related to lower intra-abdominal pressure, and improved surgical exposure. In order to safely conduct deep neuromuscular blockade, it is essential to use Sugammadex to reverse the neuromuscular block. Conventional practice is to provide moderate neuromuscular block and reverse with neostigmine. It is not possible to safely reverse deep neuromuscular block using neostogmine, as the majority of block must have worn off for neostigmine to be effective. in order to identify whether deep neuromuscular block improves quality of recovery after surgery, the investigators will conduct a randomised trial of deep versus moderate neuromuscular block, whilst minimising variance in other anaesthetic techniques and drugs used. the outcome measured will be the post-operative quality of recovery over multiple time periods using the Postoperative Quality of Recovery Scale (PostopQRS). 350 patients will be enrolled over 4 centres.

DETAILED DESCRIPTION:
Objectives

1. To identify whether the rate/quality of recovery is affected by deep neuromuscular block (DNB) and reversal with sugammadex versus light/moderate neuromuscular block reversed with neostigmine and couple with desflurane or sevoflurane in patients undergoing operative gynecological or abdominal laparoscopic surgery of at least 1-hour duration.

Hypothesis

1. The technique of deep neuromuscular block and reversal with sugammadex will result in improved quality of recovery, including cognition, compared to the current standard of care technique using light/moderate neuromuscular block reversed with neostigmine in patients undergoing operative gynecological or abdominal laparoscopic surgery of at least 1-hour duration.

Background:

Importance and assessment of quality of recovery

Recovery following general anesthesia is a complex issue confounded by the type of surgery, inflammation, different anesthetic drugs and techniques, patient co-morbidities, and differing patient and clinician perceptions of what constitutes good recovery.

Recovery is not a single entity but rather covers many aspects or domains such as physiological recovery, pain and nausea, emotion and mood, return to normal life or work activities, and cognitive function. It is an entity that is difficult to quantify, which then makes it difficult to study in a systematic manner. For anesthesiologists, poor recovery is often relayed by the surgeon days or weeks after the event, and it is usually categorized as an adverse outcome.

Research tools such as the Aldrete or the QoR scales, focus on early physiological recovery, or the immediate perioperative period. These recovery scores are not sensitive enough to measure the rate of recovery (change over time), and have not been designed for repeated measures. They are also inadequate to identify poor cognitive recovery.

In 2007, an international group of anesthesiologists and neuropsychologists formed an advisory board to create a new quality of recovery scale. The aim was to produce a tool that was simple to perform, but sensitive enough to detect change in multiple domains of recovery over time. The initial validation experiment included over 700 patients, and this work has been published in Anesthesiology. It is called the Postoperative Quality Recovery Scale (PostopQRS). Six domains of recovery are identified: physiological, nociceptive (pain and nausea) emotive (anxiety and depression), functional recovery (return of activities of daily living), cognitive recovery, and an overall patient perspective domain including satisfaction. The scale is completed prior to surgery to provide baseline values, and then repeated at user-defined intervals. From some of the subsequent discriminant validation studies, time points have included early and late measures such as 15 minutes, 40 minutes, 1 and 3 days, and 3 months after the completion of anesthesia (typically defined as after the last surgical stimulation). Recovery is broadly defined as return to baseline values or better, except for the cognitive domain where a tolerance factor is included to allow for normal performance variability, such that patients are allowed to perform a little worse than baseline as still be scored as recovered. Because repeated tests tend to have a learning effect, the cognitive domain uses parallel forms, and only a small learning has been shown.

One of the most important benefits of the PostopQRS scale is that it enables recovery to be quantified and measured. This makes it possible to compare different interventions with the express purpose of developing clinical interventions to improve quality of recovery. The PostopQRS offers a tool to provide the recovery process to be examined. There are no other tools in existence that provide a comprehensive, sensitive assessment of the multiple aspects or domains of recovery, and is yet relatively simple to perform. Validation studies have been performed and show good discriminative ability (5-8). Ease of use is facilitated by using a web based data entry system and the ability to use the telephone to conduct surveys after discharge form hospital. Telephone survey has been shown to be equivalent to face to face interviews using the PostopQRS. Further, the PostopQRS allows users to drill down to identify which recovery domain is affected for individuals in real time as well as for group audit.

Quality of recovery after operative laparoscopy

The majority of the literature compares different operative techniques with outcome measures aimed at specific complications or length of stay. Few studies include quality of recovery or quality of life measures as secondary endpoints. However, for potential benefits relating to the use of sugammadex, there are a few studies primarily centered around deep neuromuscular block (DNB) facilitating low intraabdominal inflation pressures. Most outcomes relate to operative conditions with little data on patient centered outcomes especially after discharge. The inclusion of sugammadex is to permit the use of DNB, and most comparative groups (of moderate block) are reversed with neostigmine.

It has been shown that more patients can be operated on with low intraabdominal pressure with DNB, and that operative conditions are rated as better in more patients with DNB, though it is not absolute and there are frequent crossovers. That is, there are patients with moderate block and low pressure, and equally patients with DNB requiring high inflation pressures. The very few data on patient centered outcomes show reduced pain and nausea after DNB, but lack of evidence of benefit for other recovery outcomes. This paucity of data has been stressed by review articles and editorials that DNB is associated with a modest effect on improving operating conditions but very little data to identify recovery benefits.

Sugammadex is an effective drug to reduce deep neuromuscular blockade

There is no clinical question that sugammadex is highly effective in reversing neuromuscular blockade with rocuronium or vecuronium. This has been the subject of a Cochrane review which included 18 randomized trials, showing that sugammadex can reverse blockade with rocuronium or vecuronium independent on the depth of block, and superiority to neostigmine. This aspect of sugammadex does not require further study. This translates to a low incidence of residual blockade in the PACU compared to neostigmine reversal. The "safety" benefit to using sugammadex has been proven, but this does not necessarily translate into better outcomes. Sugammadex, however, is an enabling drug to facilitate deep neuromuscular blockade, allowing the anesthesiologist to continue that block until the end of surgery and reliably reverse the block. This is just not possible with neostigmine reversal, as one must wait until a train of four count of at least 2 twitches (or TOF ratio > 0.7) to safely reverse the block with neostigmine.

Sugammadex is not a single intervention

The role of sugammadex as a single intervention can only be applied when reversing neuromuscular block, when the block is moderate and a TOF 0.7 is achieved, with the outcome restricted to reversal of blockade.

When sugammadex is used as a tool to facilitate deep muscular block, the intervention is principally the DNB rather than sugammadex. In any randomized trial comparing sugammadex with neostigmine for reversal of DNB, the extra time that anesthesia is continued in the neostigmine group will be a confounder on post-operative outcomes. In a study comparing sugammadex vs. neostigmine to reverse DNB, the anesthetic time in the neostigmine group was almost double that of the sugammadex group (47 vs 95 min). This markedly increased anesthetic duration was due to the time taken for the TOF ratio to exceed 0.9 and facilitate safe extubation. It is therefore not possible to examine the issue of deep neuromuscular block and unbundle sugammadex from the anesthetic technique required.

Outcomes and confounders when assessing post-operative quality of recovery There are a few data assessing the impact of anesthetic drugs rather than surgical techniques or different operations on the post-operative quality recovery. It is very likely that different anesthetic drugs may independently contribute to changes in post-operative quality of recovery, over and above the use of deep neuromuscular block for laparoscopic surgery.

The two most commonly used anesthetic drugs are propofol and sevoflurane. Both are relatively short acting drugs, but have a wide variation of offset, particularly with more prolonged anesthesia, and patient factors such as morbid obesity. Desflurane is a volatile agent which is very short acting, and more importantly has highly predictable offset, which is independent of patient factors such as obesity or of operation duration. In patients receiving moderate neuromuscular block and reversal with neostigmine, the use of desflurane lead to earlier response to command and return of airway reflexed compared to sevoflurane.

The investigators research group is currently conducting research into different anesthetic techniques. Previously, the investigators studied effect of desflurane vs. propofol in patients undergoing cardiac surgery, and showed less cognitive dysfunction one week after surgery but not at three months after surgery with desflurane. The investigators have recently concluded but not published a pilot study investigating propofol sedation vs. desflurane general anesthesia to supplement spinal anesthesia for total hip replacement. The participant numbers are too small for meaningful statistical analysis, but there is a trend towards improved recovery and better cognitive recovery in the desflurane group (absolute difference 15% and OR 2.3). What is interesting, though, is that the early differences were negligible, and the trend occurred at 1 month and 3 months after surgery.

In this study, the investigators wish to primarily investigate the effect of the role of DNB, and to reduce the potential for confounding from different anesthetic techniques, we will standardize the anesthetic to use the shortest acting anesthetic bundle, and use desflurane coupled with short acting opiates and multimodal analgesia in patients undergoing operative gynecological or abdominal laparoscopic surgery of at least 1-hour duration.

Clinical significance

Quality of recovery is an emerging field within anesthesia of great importance. Although large outcome studies are very important in anesthesia, there is a changing focus from "mortality and morbidity studies", to quality of recovery. The reason is that the frequency of mortality is now very low with the result that few interventions will further reduce mortality and in any event very large numbers will be required to demonstrate any improvements in surgery and anesthesia with mortality as an outcome. However early data on the PostopQRS as well as clinical reports indicate that the quality of recovery is often poor in many patients, and yet these are not identified by the treating anesthesiologist. There are implications for the individual patient, for the practice of anesthesia, and for the community (such as safe return to work or to driving).

If providing deep neuromuscular block does lead to improved quality outcomes, then it is essential to use sugammadex to reverse the block. There may be benefits (such as cognitive recovery) that may be worsened by drugs such as neostigmine and avoidance of neostigmine may be a mechanism of improving recovery. The coupling of drugs with similar offset times may further lead to improved quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants
2. operative gynecological or abdominal surgery
3. receiving general anesthesia
4. Operation expected to exceed1 hour duration
5. Participants must speak sufficient English to answer the survey questions

Exclusion Criteria:

1. Participants undergoing diagnostic laparoscopy only
2. Participants <18 years of age
3. Current pregnancy
4. Known allergy to rocuronium, neostigmine or sugammadex, or desflurane

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Royse, MD, Principal Investigator — University of Melbourne
Locations (4):
- Australia (4):
  - Northpark Private Hospital, Bundoora, Victoria
  - Melbourne Health, Parkville, Victoria
  - The Royal Womens Hospital, Parkville, Victoria
  - Victorian Comprehensive Cancer Centre, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boggett S, Chahal R, Griffiths J, Lin J, Wang D, Williams Z, Riedel B, Bowyer A, Royse A, Royse C. A randomised controlled trial comparing deep neuromuscular blockade reversed with sugammadex with moderate neuromuscular block reversed with neostigmine. Anaesthesia. 2020 Sep;75(9):1153-1163. doi: 10.1111/anae.15094. Epub 2020 May 12. PMID 32395901

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the period from June 2017 until November 2018, 350 patients were enrolled across 4 hospital sites (100 patients from the Royal Melbourne Hospital, 98 from the Peter MacCallum Cancer Centre, 88 from the Royal Women's Hospital and 64 from North Park Private Hospital).
Pre-assignment Details: No participants were excluded from the study prior to surgical procedure
Groups:
- Moderate Neuromuscular Blockade Reversed With Neostigmine: The initial dosage of a moderate block was 0.6mg/kg of rocuronium, with repeat dosage of 0.15mg/kg given if the TOF > 2.
  Once the TOF had 2 twitches, 50mcg/kg Neostigmine coupled with 20mcg/kg of atropine or 5mcg/kg of glycopyrrolate was administered for the reversal of a moderate block with a maximum dosage of 5.0mg of neostigmine.
  Extubation occurred when the TOF = 4 with no visible fade.
- Deep Neuromuscular Blockade Reversed With Sugammadex: The initial dosage of deep block was 1.2mg/kg with repeat dosages of 0.15mg/kg until PTC ≤ 2.
  Sugammadex dosage was adjusted to body weight and PTC/TOF count at the time of reversal, and not administered until PTC at least 1. The dosage was 4mg/kg when TOF=0 and PTC ≥ 1; and 2 mg/kg if TOF ≥1.
  Extubation occurred when the TOF=4 with no visible fade.
Period: Overall Study
Arm/Group | Moderate Neuromuscular Blockade Reversed With Neostigmine | Deep Neuromuscular Blockade Reversed With Sugammadex
Started | 175 | 175
Completed | 144 | 140
Not Completed | 31 | 35
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Lost to Follow-up | 25 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Neuromuscular Blockade Reversed With Neostigmine | Deep Neuromuscular Blockade Reversed With Sugammadex | Total
Number analyzed (Participants) | 175 | 175 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (16.3) | 54.4 (15.5) | 54.5 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 79 | 181
  Male | 73 | 96 | 169
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 175 | 175 | 350
ASA Status [Count of Participants; unit: Participants] — ASA physical status classification system ASA I = healthy person ASA II = mild systemic disease ASA III = severe systemic disease Population: Missing data Moderate block = 7 Deep block = 3
  Participants
    number analyzed (Participants) | 168 | 172 | 340
    ASA I | 24 | 30 | 54
    ASA II | 99 | 104 | 203
    ASA III | 45 | 38 | 83
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body mass index
  kg/m^2 | 29.5 (6.0) | 28.8 (6.1) | 29.2 (6.0)
Education [Mean (Standard Deviation); unit: years] — Years in full-time education
  years | 13.5 (4.0) | 13.3 (3.4) | 13.4 (3.5)
Alcohol consumption [Mean (Standard Deviation); unit: units/week] — Standard units consumed per week
  units/week | 4.8 (8.1) | 3.9 (6.3) | 4.3 (7.2)
Previous smoker [Count of Participants; unit: Participants] | 85 | 86 | 171
Current Smoker [Count of Participants; unit: Participants] | 24 | 15 | 39
Employment [Count of Participants; unit: Participants] — Currently employed
  Participants | 93 | 114 | 207
Surgical access [Count of Participants; unit: Participants]
  Laparoscopic surgery | 125 | 131 | 256
  Robotic-assisted | 50 | 44 | 94
Out-patient [Count of Participants; unit: Participants] | 12 | 13 | 25
Anaesthetic technique [Count of Participants; unit: Participants]
  General anaesthesia | 164 | 164 | 328
  Spinal anaesthesia | 11 | 9 | 20
  Regional block | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Recovered Cognitively at 1 Week
Description: The primary outcome will be the cognitive domain at 1 week after surgery, when it is expected that most of the acute inflammation will have resolved, and analgesia requirements minimal.
Time Frame: 1 week
Population: There were 31 participants who did not complete the cognitive assessment at 1 week in the moderate neuromuscular blockade group, whereas there were 35 participants who did not complete the cognitive assessment at 1 week in the deep neuromuscular blockade group
Measure: Number; unit: percentage of patients recovered
Arm/Group | Moderate Neuromuscular Blockade Reversed With Neostigmine | Deep Neuromuscular Blockade Reversed With Sugammadex
Number analyzed (Participants) | 144 | 140
percentage of patients recovered | 91.8 | 92.9

2. Secondary Outcome: Percentage of Patients Recovered in All Domains of the Postoperative Quality of Recovery Scale at 3 Months After the Operation
Description: Recovery for all domains and within domains of the PostopQRS scale at the other time points of measurement (15 minutes, 40 minutes 1 day, 3 days, 1 and 2 weeks, and 3 months following cessation of anesthesia). The domains of recovery are physiological, nociceptive, emotive activities of daily living, cognitive and overall patient perspective.
Time Frame: 3 months
Population: Recovery in all domains of the Postoperative Quality of Recovery Scale at 3 months after the operation
Measure: Number; unit: percentage of patients recovered
Arm/Group | Moderate Neuromuscular Blockade Reversed With Neostigmine | Deep Neuromuscular Blockade Reversed With Sugammadex
Number analyzed (Participants) | 175 | 175
percentage of patients recovered | 75.7 | 73

3. Secondary Outcome: Number of Participants With Full Reversal of Neuromuscular Blockade Prior to Extubation
Description: Compliance with protocol to ensure deep block or light/moderate block, using the train of four ratio and post tetanic count
Time Frame: 6 hours
Population: Full reversal prior to extubation (4 twitches and TOF ratio >0.9)
Measure: Number; unit: participants
Arm/Group | Moderate Neuromuscular Blockade Reversed With Neostigmine | Deep Neuromuscular Blockade Reversed With Sugammadex
Number analyzed (Participants) | 175 | 175
participants | 158 | 161

4. Secondary Outcome: Duration of Anesthesia From Induction to Cessation of the Anesthetic
Description: Duration of Anesthesia from induction to cessation of the anesthetic up to 6 hours
Time Frame: Up to 6 hours
Population: Duration of Anesthesia from induction to cessation of the anesthetic
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Moderate Neuromuscular Blockade Reversed With Neostigmine | Deep Neuromuscular Blockade Reversed With Sugammadex
Number analyzed (Participants) | 175 | 175
minutes | 165.4 (88.8) | 164 (96)

5. Secondary Outcome: Number of Participants Categorized by Level of Surgical Satisfaction
Description: Overall surgical satisfaction using a 1-5 Likert scale (1 = very unacceptable, 2 = unacceptable, 3 = acceptable, 4 = good, 5 = excellent).
Time Frame: 2 hours
Population: Surgical operating conditions
Measure: Number; unit: participants
Arm/Group | Moderate Neuromuscular Blockade Reversed With Neostigmine | Deep Neuromuscular Blockade Reversed With Sugammadex
Number analyzed (Participants) | 166 | 165
participants
  Excellent | 104 | 94
  Good | 38 | 48
  Acceptable | 20 | 16
  Unacceptable | 3 | 1
  Very Unacceptable | 1 | 1

6. Secondary Outcome: Duration of Hospital Length of Stay
Description: Duration of hospital length of stay following their procedure until hospital discharge
Time Frame: 3 days
Population: Duration of hospital length of stay following their procedure until hospital discharge
Measure: Mean (Standard Deviation); unit: days
Groups:
- Moderate Neuromuscular Blockade Reversed With Neostigmine: Moderate Neuromuscular block: participants will receive moderate neuromuscular blockade with rocuronium aiming for TOF 0-2 twitches, with neostigmine reversal when the TOF at least 3 twitches. The depth of neuromuscular block may be reduced after completion of the majority of surgical excision to TOF 3 or more
  Neostigmine
  Neostigmine: Neostigmine 50 micrograms/kg coupled with atropine 20 micrograms/kg or glycopyrrolate 5 micrograms/kg, to a maximum dose of neostigmine of 5.0 mg. The neostigmine should not be administered until the TOF has at least 3 twitches present.
- Deep Neuromuscular Blockade Reversed With Sugammadex: Deep Neuromuscular block: participants will receive DNB aiming for a post tetanic count of 1-2, which will be maintained until removal of the laparoscopic ports, with reversal using sugammadex
  Sugammadex: Reversal of neuromuscular block Sugammadex dosage will be adjusted to body weight and PTC/TOF count at the time of reversal, and not administered until PTC at least 1. Dosage will be 4mg/kg if TOF = 0 and PTC ≥ 1; and 2 mg/kg if TOF ≥1.
Arm/Group | Moderate Neuromuscular Blockade Reversed With Neostigmine | Deep Neuromuscular Blockade Reversed With Sugammadex
Number analyzed (Participants) | 175 | 175
days | 2.6 (3.5) | 1.8 (1.9)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Moderate Neuromuscular Blockade Reversed With Neostigmine | Deep Neuromuscular Blockade Reversed With Sugammadex
All-Cause Mortality (participants affected / at risk) | 0/175 | 0/175
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/175
Other Adverse Events (participants affected / at risk) | 0/175 | 0/175

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT03034577/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT03034577/SAP_001.pdf